CLINICAL TRIAL: NCT01502111
Title: Improved Knowledge Through Better Data, Implementing and Evaluating a Novel Consensus-based Template for Uniform Reporting of Data From Pre-hospital Airway Management - a Prospective Multicentre Observational Study
Brief Title: Airway Management Study in Physician Manned Helicopter Emergency Medical Services
Acronym: AIRPORT
Status: Completed | Type: Observational
Sponsor: Norwegian Air Ambulance Foundation (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NLA-3104-01/02
Record Dates: First submitted 2011-12-22; First posted 2011-12-30 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Trauma; Cardiac Arrest; Emergencies
Keywords: decreased level of consciousness; hypoxemia; ineffective ventilation; airway obstruction; combative or unresponsive; relief of pain or distress; cardiopulmonary arrest
MeSH Terms: conditions — Wounds and Injuries; Heart Arrest; Emergencies; Hypoxia; Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Airway management: Patients receiving advanced airway management in physician manned helicopter emergency medical services over a 12-month period.

SUMMARY:
An international airway management expert group has recently developed an Utstein-style template for uniform reporting of data from prehospital advanced airway management. Implementing and validating the template will result in a high quality dataset and allow for research cooperation and comparison of airway management practice between EMS systems, and across different patient populations. Such a dataset will hopefully contribute to new knowledge in the field of prehospital advanced airway management.

DETAILED DESCRIPTION:
Advanced airway management and ventilatory control is generally regarded as vital in the management of seriously ill or injured patients, and can be critical interventions in patients with out-of-hospital emergencies. However, interventions like endotracheal intubation suffer from lack of clear evidence of a beneficial effect. Despite the publication of numerous airway management studies, inconsistent and imprecise reporting of data across heterogenous patient populations and EMS systems persists. The questions of how, and by whom, pre-hospital advanced airway management should be performed remains disputed.

Several authors have proposed appropriate guidelines and algorithms for management of prehospital airway and difficult intubation. The guidelines emphasize the importance of promoting patient safety and avoiding errors, and also recognise the importance of rescuers level of airway skills competence. Drug-assisted rapid sequence intubation (RSI) is an important, but potentially harmful, component of prehospital advanced airway management in EMS services. Even physicians working in the prehospital scene may find it challenging to maintain an adequate level of advanced airway competence in order to stay proficient. Better training methods and systems are warranted.

The recognition of endotracheal intubation as a "complex intervention" marks the need for an international standard for documenting and reporting data from prehospital intubations in severely injured or ill patients, alongside a standardization of research data collection to eliminate confounding factors. An international airway management expert group has recently developed an Utstein-style template for uniform reporting of data from prehospital advanced airway management. Implementing and validating the template will result in a high quality dataset and allow for research cooperation and comparison of airway management practice between EMS systems, and across different patient populations. Such a dataset will hopefully contribute to new knowledge in the field of prehospital advanced airway management.

The specific aims for the first two studies in this project are defined as follows:

1. Describe the characteristics and outcome of advanced prehospital airway management in Helicopter Emergency Medical Services (HEMS) that provide the full range of advanced emergency airway management.
2. Identify which groups of critically injured or ill patients will benefit most from competent advanced prehospital airway management, and identify specific areas for future research.

In this multicentre study, we have enlisted 21 key international HEMS services from 6 countries (UK, Australia, Hungary, Finland, Switzerland and Norway), and will collect data according to the Utstein style template over a 12 month study period starting January 1, 2012.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring and receiving prehospital advanced airway management on HEMS primary missions.
* Advanced airway management is defined as the attempted insertion of an advanced airway adjunct (including endotracheal intubation, alternative airways, and surgical airway /cricothyroidectomy) or the administration of ventilatory assistance/support (including bag-mask ventilation-BMV, BIPAP/CPAP or other ventilatory support).
* Advanced prehospital advanced airway management is further defined as any airway management beyond manual opening of the airway and use of simple airway adjuncts, such as a Guedel airway or supplemental oxygen

Exclusion Criteria:

* Patients receiving advanced airway management during so-called secondary missions (or inter-hospital transfer).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving advanced airway management in physician manned helicopter emergency medical services over a 12-month period.
  Data reported according to the Utstein style template for uniform reporting of data from prehospital advanced airway management
Sampling Method: Probability Sample
Enrollment: 2333 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who survive to hospital admission | Time from injury/illness to admission hospital, up to 24 hours

SECONDARY OUTCOMES:
Number of participants with adverse events during airway interventions | Time from injury/illness to admission hospital, up to 24 hours
  Airway intervention success rates and airway management related complications. We will calculate airway intervention success rates, frequency and complications for the entire cohort and for key subsets (like cardiac arrest, medical, trauma, pediatric patients and RSI/alternative airways), population demographics and prevalence of adverse effects (like missed intubations, bradycardia, hypotension, hypoxia). Outcome and patient characteristics will be analysed and described.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sollid, MD, PhD, Study Chair — Norwegian Air Ambulance Foundation; Geir A Sunde, MD, Principal Investigator — Norwegian Air Ambulance Foundation
Locations (1):
- Department of Research and Development, Norwegian Air Ambulance Foundation, Drøbak, Drøbak, Norway

REFERENCES:
- [Derived] Sunde GA, Sandberg M, Lyon R, Fredriksen K, Burns B, Hufthammer KO, Roislien J, Soti A, Jantti H, Lockey D, Heltne JK, Sollid SJM. Hypoxia and hypotension in patients intubated by physician staffed helicopter emergency medical services - a prospective observational multi-centre study. BMC Emerg Med. 2017 Jul 11;17(1):22. doi: 10.1186/s12873-017-0134-5. PMID 28693491
- [Derived] Sunde GA, Heltne JK, Lockey D, Burns B, Sandberg M, Fredriksen K, Hufthammer KO, Soti A, Lyon R, Jantti H, Kamarainen A, Reid BO, Silfvast T, Harm F, Sollid SJ; Airport Study Group. Airway management by physician-staffed Helicopter Emergency Medical Services - a prospective, multicentre, observational study of 2,327 patients. Scand J Trauma Resusc Emerg Med. 2015 Aug 7;23:57. doi: 10.1186/s13049-015-0136-9. PMID 26250700